CLINICAL TRIAL: NCT03955094
Title: Clinical Evaluation of Ambu® Auragain™ as a Conduit for Intubation in Paediatrics
Brief Title: Ambu® Auragain™ as a Conduit for Intubation in Paediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Lim Su Sian, Medical officer UD 48, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Auragain study
Record Dates: First submitted 2019-05-08; First posted 2019-05-17 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Pediatric Endotracheal Intubation
Keywords: AMBU® AURAGAIN™; intubation in paediatrics; flexible scope guided intubation; success rate of intubation; glottic view; supraglottic airway intubation; efficacy safety

STUDY DESIGN:
Intervention Model Description: Prospective observational study All eligible patients will be approached and recruited All patients will be assigned to a single group - the use of AMBU® AURAGAIN™ as a conduit for flexible scope intubation No comparison groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMBU® AURAGAIN™ device (Experimental): Assess feasibility of AMBU® AURAGAIN™ as an intubating device in paediatrics
  Interventions: Device: Intubation via AMBU® AURAGAIN™

INTERVENTIONS:
Device: Intubation via AMBU® AURAGAIN™ — Success rate of paediatric intubation through AMBU® AURAGAIN™
  Other Names: AMBU® AURAGAIN™; Supraglottic device

SUMMARY:
This study will be conducted as a prospective observational study

This study will be done in any of the operating theatres of University Malaya Medical Centre

This study will involve paediatric cases ( ages 3-12 years )posted for elective operations which require general anaesthesia with endotracheal intubation

Ambu Aura Gain will be used as a conduit for intubation

DETAILED DESCRIPTION:
All eligible participants will be approached and recruited Informed consent will be obtained Induction of general anesthesia will be as per usual standardized method Ambu® Auragain™ will be inserted A paediatric flexible endoscope will be used to view the glottis and railroad an endotracheal tube into the trachea Placement is confirmed and number of attempts and time required for successful intubation is recorded Ambu® Auragain™ will be removed Number of attempts and time taken for removal of Ambu® Auragain™ will be recorded Any complications will be noted and recorded

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients aged 3 - 12 years old
* American Society of Anaesthesiologist (ASA) 1-2 patients
* Patients must require standard endotracheal intubation for the procedure posted

Exclusion Criteria:

* Documented history of difficult airway in previous general anaesthesia
* Clinical features of difficult airway on physical examination
* Syndromic patients, facial deformities, dental deformities, patients with facial trauma
* Patients with recent (less than 2 weeks) or ongoing upper respiratory tract infection
* Patients with existing pulmonary diseases or any risk of bronchospasm
* Patients with known gastric outlet obstruction, reflux disease, or any risk of aspiration
* Any other contraindication for device placement
* Operations requiring specialised endotracheal tubes
* Emergency operations or unanticipated difficult airway cases
* Refusal of parental informed consent

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Time taken to successful intubation via the Ambu® AuraGain™ | Time taken during procedure ( measured in seconds )
  Successful intubation is confirmed via the equal air entry heard bilaterally on auscultation and a positive capnograph tracing

SECONDARY OUTCOMES:
Time taken required for removal of Ambu® AuraGain™ post intubation | Time taken during procedure ( measured in seconds )
  Successful removal of device is confirmed by equal air entry heard bilaterally on auscultation and a positive capnograph tracing

OTHER OUTCOMES:
Time required for insertion of Ambu® AuraGain™ | Time taken during procedure ( measured in seconds )
  Device insertion is limited to two attempts
Determine oropharyngeal leak pressure of Ambu® AuraGain™ | Immediately post procedure- insertion of Ambu® AuraGain™ ( measured in mmHg )
  Standard oropharyngeal leak test performed

CONTACTS AND LOCATIONS:
Overall Officials: Ismiarti S Ina, MAnaes(UM), Study Chair — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinha R, Chandralekha, Ray BR. Evaluation of air-Q intubating laryngeal airway as a conduit for tracheal intubation in infants--a pilot study. Paediatr Anaesth. 2012 Feb;22(2):156-60. doi: 10.1111/j.1460-9592.2011.03710.x. PMID 21973052
- [Background] Pandey RK, Subramanium RK, Darlong V, Lekha C, Garg R, Punj J, Rewari V, Bajpai M. Evaluation of glottic view through Air-Q Intubating Laryngeal Airway in the supine and lateral position and assessing it as a conduit for blind endotracheal intubation in children in the supine position. Paediatr Anaesth. 2015 Dec;25(12):1241-7. doi: 10.1111/pan.12746. Epub 2015 Sep 29. PMID 26417722
- [Background] Jagannathan N, Kozlowski RJ, Sohn LE, Langen KE, Roth AG, Mukherji II, Kho MF, Suresh S. A clinical evaluation of the intubating laryngeal airway as a conduit for tracheal intubation in children. Anesth Analg. 2011 Jan;112(1):176-82. doi: 10.1213/ANE.0b013e3181fe0408. Epub 2010 Nov 16. PMID 21081777
- [Background] Jagannathan N, Sohn LE, Sawardekar A, Gordon J, Shah RD, Mukherji II, Roth AG, Suresh S. A randomized trial comparing the Ambu (R) Aura-i with the air-Q intubating laryngeal airway as conduits for tracheal intubation in children. Paediatr Anaesth. 2012 Dec;22(12):1197-204. doi: 10.1111/pan.12024. Epub 2012 Sep 13. PMID 22971118
- [Background] Jagannathan N, Sohn L, Ramsey M, Huang A, Sawardekar A, Sequera-Ramos L, Kromrey L, De Oliveira GS. A randomized comparison between the i-gel and the air-Q supraglottic airways when used by anesthesiology trainees as conduits for tracheal intubation in children. Can J Anaesth. 2015 Jun;62(6):587-94. doi: 10.1007/s12630-014-0304-9. Epub 2014 Dec 24. PMID 25537736
- [Background] Girgis KK, Youssef MM, ElZayyat NS. Comparison of the air-Q intubating laryngeal airway and the cobra perilaryngeal airway as conduits for fiber optic-guided intubation in pediatric patients. Saudi J Anaesth. 2014 Oct;8(4):470-6. doi: 10.4103/1658-354X.140841. PMID 25422603